CLINICAL TRIAL: NCT04505501
Title: Reducing HIV Persistence in Lymph Nodes by Interleukin-15 (IL-15) Receptor Super-agonist (N-803) in Individuals With Acute HIV Infection
Brief Title: Reducing HIV Persistence in Lymph Nodes by Interleukin-15 (IL-15) Receptor Super-agonist (N-803) in Acute HIV Infection
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Thai Red Cross AIDS Research Centre (Other)
Collaborators: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other); Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RV550
Record Dates: First submitted 2020-07-13; First posted 2020-08-10 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: HIV/AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — ALT-803

STUDY DESIGN:
Masking Description: This study is unblinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- N-803 (Experimental): Step 1: N-803 at 6mcg/kg every 3 weeks for 3 doses plus ART (n=10) Step 2 : N-803 at 6mcg/kg at week 0 single dose (n=8), ATI after N-803 injection until week 12 (If meet criteria to restart ART, participants will go to step 3).
  Step 3: ART restart (week 0 to week 12).
  Interventions: Drug: N-803
- Control (No Intervention): Step 1: ART alone (n=5) Step 2 : N-803 at 6mcg/kg at week 0 single dose (n=8), ATI after N-803 injection until week 12 (If meet criteria to restart ART, participants will go to step 3).
  Step 3: ART restart (week 0 to week 12).

INTERVENTIONS:
Drug: N-803 — N-803 is a novel IL-15 superagonist complex that enhances NK cell and CD8+ T-cell proliferation and activation.
  Other Names: ALT-803
  Arms: N-803

SUMMARY:
Reducing HIV persistence in lymph nodes by Interleukin-15 (IL-15) Receptor super-agonist (N-803) in Individuals with Acute HIV Infection

DETAILED DESCRIPTION:
This is a phase II, randomized, unblinded, controlled trial to investigate the safety, tolerability and immunomodulation effect of combining N-803 with ART during AHI. The study will be conducted at the Thai Red Cross AIDS Research Centre (TRCARC)/King Chulalongkorn Memorial Hospital and the Faculty of Medicine, Chulalongkorn University in Bangkok, Thailand.

Eligible participants will be asked to undergo LN Bx at baseline (untreated AHI), prior to initiating dolutegravir-based ART.

This study will have three steps.

In Step 1, N-803 will be administered subcutaneously at weeks 0, 3, 6 (total 3 doses) and will be initiated together with ART. Participants will be asked to undergo a second inguinal LN Bx on the opposite groin approximately at week 6 (no later than 1 week after completion of study agents). They will be followed for safety parameters at weeks 8 and 12, after which they will roll over to the RV412, WRAIR#2178 safety monitoring protocol. Step 1 duration for individual participants will be approximately 12 weeks. Step 1 has been completed as per protocol by 12 participants, 8 N-803 recipients and 4 ART only participants and study recruitment has ended.

In Step 2, participants who have completed Step 1 as per protocol and remain virologically controlled will be given a single dose of N-803 followed by ATI. The N-803 dose will be offered to all these participants regardless of initial randomization in Step 1. In Step 2, N-803 will be administered at Step 2 week 0 followed by ATI on the same day. The participants will be followed during ATI for viral rebound and monitored for the restart criteria for a maximum of 12 weeks. Participants who do not meet ART restart criteria at the end of Step 2 will proceed to RV412, WRAIR#2178 for safety follow-up.

In Step 3, participants who did restart ART during Step 2 will be monitored for safety after restarting ART. Participants will be monitored every 2 weeks for a total of 12 weeks in Step 3. Any participants who may not have achieved HIV suppression by the end of Step 3 and the study will also proceed to RV412, WRAIR#2178 for continuing safety follow-up. Total study duration through data analysis and closure is estimated at five years.

It is hypothesized that N-803 initiated with ART during AHI, will be safe, and will lead to a reduction of HIV reservoir size in LN, demonstrated by decreased frequencies of vRNA+ and vDNA+ cells in the LNs, in comparison with ART alone.

ELIGIBILITY:
Inclusion Criteria for step 1:

1. Age 18 years and above.
2. Acute HIV infection (Fiebig I to V: Fiebig I: RNA+, p24 antigen-; Fiebig II: p24 antigen+, IgM-; Fiebig III: IgM+, Western Blot-; Fiebig IV: Western Blot indeterminate; Fiebig V: Western Blot+ without p31 protein band)
3. All female participants of childbearing potential must have a negative urine pregnancy test at the screening visit
4. Women of child bearing potential and men with partners of child bearing potential must agree to use effective contraception (as defined in section 8.1.2 Pregnancy Risks) during therapy and for 4 months after completion of therapy
5. Can read and write Thai and/or English language and must be able to understand and complete the informed consent process
6. Must successfully complete a Test of Understanding (TOU) prior to enrollment as described in Section 7.1
7. Willing to undergo inguinal LN Bx at two time points (baseline and week 6) and blood draws during each study visit
8. Willing to participate for the duration of the study visits and follow up.

Exclusion Criteria for step 1:

1. Pregnant, breastfeeding, or unwilling to practice birth control during participation in the study
2. Active or recent malignancy requiring systemic chemotherapy or surgery in the preceding 36 months or for whom such therapies are expected in the subsequent 12 months; minor surgical removal of localized skin cancers (squamous cell carcinoma, basal cell carcinoma) are not exclusionary
3. Receipt of any vaccine within 2 weeks prior to study enrollment and anticipated need for any vaccine within 2 weeks prior to or after any of the study agent administrations.
4. Current or anticipated use of systemic steroid medications.
5. Any clinically significant acute or chronic medical condition, including, pulmonary, hepatic, renal, gastrointestinal, genitourinary, hematological, coagulation, that in the opinion of the investigator would preclude participation (e.g., history of seizure disorders, cardiac disease, bleeding/clotting disorder, autoimmune disease, active malignancy, poorly controlled asthma, active tuberculosis or other systemic infections, etc.)
6. Chronic liver disease
7. Active and poorly controlled atherosclerotic cardiovascular disease (ASCVD), as defined by 2013 ACC/AHA guidelines, including a previous diagnosis of any of the following: (a) acute myocardial infarction, (b) acute coronary syndromes, (c) stable or unstable angina, (d) coronary or other arterial revascularization, (e) stroke, (f) transient ischemic attack, or (g) peripheral arterial disease presumed to be of atherosclerotic origin
8. History of potential immune-mediated medical conditions
9. Serious illness requiring systemic treatment and/or hospitalization in the 3 months prior to study enrollment
10. Major psychiatric illness and/or substance use during the past 12 months that in the opinion of the investigator would preclude participation
11. Concurrent treatment with immunomodulatory drugs, and/or exposure to any immunomodulatory drug in the 4 weeks prior to study enrollment
12. Exposure to any experimental therapies within 90 days of study entry
13. Pre-exposure prophylaxis (PrEP) use within 90 days of study entry

Inclusion criteria for Step 2:

1. Completed Step 1 as per protocol
2. Plasma HIV-1 RNA <50 copies/mL at the Step 2 screening visit
3. CD4 T-cell count ≥400 cells/mm3 at the Step 2 screening visit Note: The CD4 T-cell count can be repeated once, provided that the repeat is done within 1 week prior to Step 2 entry.
4. No CDC Category C event after study entry
5. Documented negative hepatitis B virus (HBV) surface antigen (HBsAg) at the screening Step 2 visit.
6. Documented negative hepatitis C virus (HCV) antibody (anti-HCV) or negative HCV RNA (if anti-HCV reactive) at the Step 2 screening visit
7. For persons of childbearing potential, negative pregnancy test at the Step 2 screening visit.
8. Persons of childbearing potential must agree to not become pregnant and use two methods of contraception if engaging in sexual activity that could lead to pregnancy. One contraceptive method must be from the list of highly effective methods listed in section 7.12. The second method of contraception must be from the barrier methods also listed in section 7.13.
9. Willingness to abstain from sexual intercourse, or use a condom, or partner(s) using pre-exposure prophylaxis consistently during ATI and until plasma HIV-1 RNA is less than limit of detection after ART restart with all partners that are HIV-uninfected or serostatus unknown.
10. Willingness to participate in ATI for up to 12 weeks.
11. Willingness to restart ART according to study guidelines.

Exclusion Criteria for Step 2 ATI

1. Virologic failure (two consecutive HIV-1 RNA >1000 copies/mL)
2. Intercurrent illness, new medical diagnosis, laboratory abnormality, sign, or symptom that, in the opinion of the site investigator, would place participant at higher risk of morbidity during ATI.
3. Receipt of any non-nucleoside reverse transcriptase inhibitor (NNRTI) within 60 days before Step 2 entry.
4. Receipt of long-acting ART such as long-acting cabotegravir (CAB LA) or long-acting rilpivirine (RPV LA) at any point after study entry.
5. Failure by the participant to attend three consecutive Step 1 study visits.
6. Pregnancy or breastfeeding.
7. Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Rate of occurrence of ≥ grade 3 adverse events determined to be related (Safety) | at time of study completion at week 12
  Rate of occurrence of ≥ grade 3 adverse events determined to be related
Frequency of vRNA+ and vDNA+ cells and levels of vDNA and vRNA in LNs | At baseline (week 0) and week 6
  Frequency of vRNA+ and vDNA+ cells and levels of vDNA and vRNA in LNs
Frequency, phenotype and function of CD8+ T cells and innate cells in LNs | At baseline (week 0) and week 6
  Frequency, phenotype and function of CD8+ T cells and innate cells in LNs
Time (days) from ATI to first documented HIV-1 RNA viral rebound of ≥1000 copies/mL following ATI. | viral rebound during Step 2 ATI
  Time (days) from ATI to first documented HIV-1 RNA viral rebound of ≥1000 copies/mL following ATI.

SECONDARY OUTCOMES:
Frequency, phenotype and function of NK, T, B and other immune cells in LNs and blood | Step 1 weeks 0, 3, 6, 12; Step 2 weeks 0, 2, 4, 6, 8, 10; Step 3 weeks 0, 2, 4, 6, 8, 10, 12
  Frequency, phenotype and function of NK, T, B and other immune cells in LNs and blood
HIV-specific antibody levels and ADCC, ADCP, ADCVI activities | Step 1 weeks 0, 3, 6, 12; Step 2 weeks 0, 2, 4, 6, 8, 10; Step 3 weeks 0, 2, 4, 6, 8, 10, 12
  HIV-specific antibody function as measured by Antibody-dependent cellular cytotoxicity (ADCC), antibody-dependent cellular phagocytosis (ADCP) and Antibody-dependent cell-mediated viral inhibition (ADCVI) levels.
Frequency of cells harboring HIV-1 vDNA, vRNA, intact genome and replication competent HIV-1 in PBMC | Step 1 weeks 0, 3, 6, 12; Step 2 week 0; Step 3 week 12
  Frequency of cells harboring HIV-1 vDNA, vRNA, intact genome and replication competent HIV-1 in PBMC
Host and viral genes by transcriptome analysis | Step 1 week 0 and 6
  Host and viral genes by transcriptome analysis
Immune activation markers in blood | Step 1 weeks 0, 3, 6, 12; Step 2 weeks 0, 2, 4, 6, 8, 10; Step 3 weeks 0, 2, 4, 6, 8, 10, 12
  Immune activation markers in blood
Immune activation markers in CSF | Step 1 week 0, 6; Step 2 week 0; Step 3 week 0, 12
  Immune activation markers in CSF
Extent of cerebral inflammation in MR Spectroscopy (MRS) | Step 1 week 0, 6; Step 2 week 0; Step 3 week 0, 12
  Extent of cerebral inflammation in MR Spectroscopy (MRS)
Viral load area under the curve (AUCv) | during the 4 weeks after viral rebound
  Viral load area under the curve (AUCv)
Responses to pilot discrete choice experiment survey | Step2 wk0
  Describe participant preferences about participation in HIV remission trials with treatment interruptions

CONTACTS AND LOCATIONS:
Overall Officials: Sandhya C Vasan, MD PhD, Study Chair — Henry M. Jackson Foundation for the Advancement of Military Medicine
Locations (1):
- Thai Red Cross AIDS Research Centre, Bangkok, Bangkok, Thailand